CLINICAL TRIAL: NCT06945744
Title: Carbohydrate Counting /Bolus Calculator Mobile Application Improves Time in Range in Adults With Type 1 Diabetes Subjects
Brief Title: Carbohydrate Counting and Bolus Calculator Mobile Application Improves Time in Range in Adults With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Fahad Medical City (Other Government)
Responsible Party: Principal Investigator, Sara Albabtain, Senior Clinical Dietitian, King Fahad Medical City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-630; 023-015 (Other Grant/Funding Number: King Fahd Medical City)
Record Dates: First submitted 2025-03-15; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus, Type I
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: A 12-week randomized controlled trial was conducted at King Fahad Medical City. Participants with T1DM who were using multiple insulin injections and Libre flash glucose monitors were randomly assigned to either CHOC-BC intervention (n = 64) or control (n = 63) group to perform conventional treatment. The primary endpoint was the time in range (TIR; 70-180 mg/dL).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participants receiving standard diabetes education (Active Comparator): The control group received a standard diabetic educational diet plan emphasizing regular meal timing and distribution. This plan included three main meals and 2-3 snacks daily while encouraging the avoidance of high glycemic and high-fat foods.
  Interventions: Other: Standard Treatment
- Participants using the Carbohydrate Counting/Bolus Calculator Mobile Application (Experimental): Eligible participants provided informed consent and underwent baseline assessments, including demographics, medical history, insulin doses, and fasting blood samples for HbA1c and lipid profile. Participants used the FreeStyle Libre 2 sensor, with AGP data collected bimonthly. The primary outcome was Time in Range (TIR, 70-180 mg/dL), while secondary outcomes included TAR, TBR, GV%, GMI, HbA1c, and BMI.
  A registered dietitian provided structured CHOC-BC education. The intervention group used the CHOC-BC app, validated against expert-calculated carbohydrate counts, while the control group followed standard diabetes education. Virtual follow-ups occurred bimonthly for three months. At study completion, HbA1c, lipid profile, insulin doses, weight, and AGP data were collected for comparison.
  Interventions: Device: Carbohydrate

INTERVENTIONS:
Other: Standard Treatment — The control group followed a standard diabetic habitual diet
  Arms: Participants receiving standard diabetes education
Device: Carbohydrate — Eligible participants provided informed consent and underwent baseline assessments, including demographics, medical history, insulin doses, and fasting blood samples for HbA1c and lipid profile. Participants used the FreeStyle Libre 2 sensor, with AGP data collected bimonthly. The primary outcome was Time in Range (TIR, 70-180 mg/dL), while secondary outcomes included TAR, TBR, GV%, GMI, HbA1c, and BMI.
  A registered dietitian provided structured CHOC-BC education. The intervention group used the CHOC-BC app, validated against expert-calculated carbohydrate counts, while the control group followed standard diabetes education. Virtual follow-ups occurred bimonthly for three months. At study completion, HbA1c, lipid profile, insulin doses, weight, and AGP data were collected for comparison.
  Arms: Participants using the Carbohydrate Counting/Bolus Calculator Mobile Application

SUMMARY:
Introduction: Accurate insulin bolusing requires advanced knowledge of carbohydrate counting and correction doses, which can be supported by mobile technology.

Objective: To evaluate the effectiveness and safety of a mobile application for carbohydrate counting and bolus calculation (CHOC-BC) in adults with type 1 diabetes mellitus (T1DM).

Methods: This is a 12-week randomized controlled trial conducted at King Fahad Medical City. Adults with T1DM using multiple daily insulin injections and Libre flash glucose monitoring systems are randomly assigned to either the CHOC-BC intervention group or a control group receiving conventional treatment. The primary endpoint is the time in range (TIR; 70-180 mg/dL).

DETAILED DESCRIPTION:
This is a single-center, randomized, controlled trial evaluating the effectiveness of a mobile application, CHOC-BC, designed to assist adults with type 1 diabetes mellitus (T1DM) in carbohydrate counting and insulin bolus calculation.

The study is conducted at King Fahad Medical City over a 12-week period. Participants are randomized into two groups: the intervention group uses the CHOC-BC mobile app, while the control group continues with standard diabetes management practices.

Participants are required to use flash glucose monitoring systems and multiple daily insulin injections. The primary outcome is the percentage of time that glucose levels remain within the target range (70-180 mg/dL), assessed using continuous glucose data. Secondary outcomes include time spent in hypoglycemia and hyperglycemia, changes in body weight, and user engagement with the application.

The study seeks to determine whether digital support tools can improve glycemic outcomes and simplify self-management among adults with T1DM.

ELIGIBILITY:
Inclusion Criteria:

Male or female participants aged 18-60 years Clinical diagnosis of type 1 diabetes mellitus (T1DM) for at least one year HbA1c >6.5% (48 mmol/mol) Using multiple daily insulin injections as the method of T1DM treatment Basic knowledge of carbohydrate counting (CHOC) Regular use of a smartphone operating on iOS 13 or higher or Android 11 Active users of the Libre 2 flash glucose monitoring system Sensor capture rate greater than 30%

Exclusion Criteria:

Limited literacy Use of an insulin pump Pregnant or breastfeeding Diagnosed with ischemic heart disease Presence of multiple comorbidities where low glucose levels may pose a risk Unwillingness or inability to comply with the study protocol Following a very low-carbohydrate diet (<10% of daily intake from carbohydrates)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2023-05-21 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Time in Range 70-180 mg/dl | From enrollment to the end of treatment at 12 weeks
  Percentage of time that glucose levels are within the target range (70-180 mg/dL) as measured by continuous glucose monitoring (CGM). TIR will be assessed at baseline and after the 12-week intervention period.

SECONDARY OUTCOMES:
Percentage of Time with Glucose >250 mg/dL | From enrollment to the end of treatment at 12 weeks
  Percentage of time that glucose levels exceed 250 mg/dL as measured by continuous glucose monitoring (CGM). This measure is used to assess the duration of hyperglycemia during the study period.
Coefficient of Variation of Glucose Levels | From enrollment to the end of treatment at 12 weeks
  Glucose variability (GV) will be assessed using standard deviation and coefficient of variation derived from continuous glucose monitoring data. This outcome measures the degree of glucose fluctuations throughout the study period.
Average Glucose Level Based on CGM Data | From enrollment to the end of treatment at 12 weeks
  Mean glucose levels will be calculated using CGM data collected over the 12-week study period. This outcome reflects average blood glucose concentration over time.

OTHER OUTCOMES:
Bi-Monthly Time in Range (70-180 mg/dL) from CGM | From enrollment to the end of treatment at 12 weeks
  To monitor safety and trend responses over time, time in range (TIR; 70-180 mg/dL) will be assessed every 2 weeks in the intervention group using continuous glucose monitoring. This will help identify short-term changes during the course of the 12-week intervention.
Time Spent Below 70 mg/dL, Number of Hypoglycemia Events, and Changes in Weight/BMI [Safety] | From enrollment to the end of treatment at 12 weeks
  Safety will be evaluated through CGM data on hypoglycemia, including time spent with glucose levels below 70 mg/dL and the number of low-glucose events. Weight and BMI will also be monitored throughout the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Kinf Fahad Medical City, Riyadh, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to confidentiality and data privacy concerns.

REFERENCES:
- See also: Carbohydrate Counting and bolus calculator Application — https://apps.apple.com/sa/app/ikfmc/id478245466